CLINICAL TRIAL: NCT06207955
Title: Does Intra-articular Injection of Platelet-Rich Fibrin After Arthrocentesis Followed by Lateral Pterygoid Muscle Injection With Botulinum Toxin Type A Improve Clinical Outcomes for Anterior Disc Displacement?
Brief Title: I-PRF After Arthrocentesis Plus Botox Injection to Lateral Pterygoid Muscle in Treatment of Anterior Disc Displacement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Ahmed Taha Ahmed Mohamed, Master student of oral and maxillofacial surgery, Fayoum University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 23122023
Record Dates: First submitted 2023-12-23; First posted 2024-01-17 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: TMJ Disc Disorder; TMJ Pain
Keywords: Anterior Disc Displacement; TMJ Clicking; I-PRF; Lateral Pterygoid Muscle; Arthrocentesis; Botulinum Toxin Type A
MeSH Terms: interventions — Botulinum Toxins, Type A; Arthrocentesis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TMJ arthrocentesis + (I-PRF) injection & injection of Botox to lateral pterygoid muscle (Active Comparator)
  Interventions: Drug: TMJ Arthrocentesis Followed By Injectable Platelet Rich Fibrin And Botulinum Toxin Type A
- TMJ arthrocentesis followed by intra-articular injection of liquid platelet rich fibrin ( I-PRF ) (Active Comparator)
  Interventions: Drug: TMJ Arthrocentesis Followed By Injectable Platelet Rich Fibrin
- TMJ arthrocentesis (Active Comparator)
  Interventions: Drug: TMJ Arthrocentesis

INTERVENTIONS:
Drug: TMJ Arthrocentesis Followed By Injectable Platelet Rich Fibrin And Botulinum Toxin Type A — TMJ Arthrocentesis I-PRF Intra-articular Injection Botulinum Toxin Type A to Lateral Pterygoid Muscle
  Arms: TMJ arthrocentesis + (I-PRF) injection & injection of Botox to lateral pterygoid muscle
Drug: TMJ Arthrocentesis Followed By Injectable Platelet Rich Fibrin — TMJ Arthrocentesis I-PRF Intra-articular Injection
  Arms: TMJ arthrocentesis followed by intra-articular injection of liquid platelet rich fibrin ( I-PRF )
Drug: TMJ Arthrocentesis — TMJ Arthrocentesis By Saline
  Arms: TMJ arthrocentesis

SUMMARY:
Aim of Study : To evaluate the efficacy of TMJ arhtrocentesis followed by injection of liquid platelet rich fibrin (I-PRF ) in addition to intramuscular injection of lateral pterygoid muscle with botulinum toxin on clinical outcomes of painful TMJ , maximum mouth opening , joint sounds and range of lateral movement in patients with TMJ anterior disc displacement with reduction

Hypothesis : Intramuscular injection of lateral pterygoid muscle with botulinum toxin plus TMJ intra-articular injection of liquid platelet rich fibrin after arthrocentesis are more effective than TMJ arthrocentesis followed by intra-articular injection of ( I-PRF ) or TMJ arthrocentesis only .

ELIGIBILITY:
Inclusion Criteria:

* Patients with painful tmj during jaw movements
* Patients with joint sounds ( clicking ) during jaw opening and mastication
* Patients age range from 16 years old to 45 years old
* Patients with Class I maxillo-mandibular relationship
* Patients with reduced mouth opening
* All patients diagnosed clinically and radiographically by MRI as TMJ anterior disc displacement with reduction

Exclusion Criteria:

* Patient with history of recent trauma
* Patients with malocclusion
* Patients with systematic condition that affect bone and joints such as osteoarthritis , systemic lupus and epilepsy .
* Patients allergic to botox injection
* Pregnant or lactating females
* Patients with non-reducible disc on MRI
* Patients contraindicated to exposure to MRI
* Patients with previous tmj arthrocentesis , arthroscopy or TMJ surgery
* Significant mechanical obstruction that prevents mouth opening, acute capsulitis, benign or malignant temporomandibular joint lesions.
* Patients with blood diseases, and coagulation disorders

Ages: 16 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 39 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Maximum Mouth Opening | 6 months
  Maximum mouth opening will be measured as the distance from incisal edges of the upper and lower central incisors using a ruler and will be evaluated preoperatively , immediately after the procedure , 1month , 3 months and 6 months postoperative .

SECONDARY OUTCOMES:
Clicking | 6 months
  Joint sounds also will be evaluated during opening and closing of the jaws and during lateral movements preoperatively , immediately after the procedure , 1 months , 3 months and 6 months postoperative
Lateral movement | 6 months
  Range of lateral mandibular movement will be measured using Vernier caliper in millimeters as the horizontal distance extending from maxillary midline to mandibular midline by asking the patient to move the mandible to one side then to the other side to maximum extent

IPD SHARING:
Plan to Share IPD: Undecided